CLINICAL TRIAL: NCT06141408
Title: A Community-based Intervention to Increase PrEP Initiation in Prince George's County, Maryland: Reducing HIV Stigma and Increasing Social Support
Brief Title: PrEP Intervention in Prince George's County, Maryland
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: George Mason University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GeorgeMU
Record Dates: First submitted 2023-11-10; First posted 2023-11-21 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Hiv; Mental Health Issue; Support, Family
Keywords: HIV; Stigma; Support; PrEP
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MPowerment PrEP Promotion Intervention (Experimental): This is the arm engaging in the stigma-reduction and support-increasing activities aimed to increase PrEP use.
  Interventions: Behavioral: MPowerment PrEP Promotion Intervention
- Standard of Care (No Intervention): This is the arm not engaging in the stigma-reduction and support-increasing activities. This arm will receive standard referreals to PrEP knowledge resources and providers.

INTERVENTIONS:
Behavioral: MPowerment PrEP Promotion Intervention — In-person events will focus on five specific goals: Fostering a sense of community acceptance and social connection, promoting self-acceptance of sexual identity, teaching skills for navigating healthcare, reducing PrEP stigma, and providing education on HIV risk. In accordance with the MPowerment model, In collaboration with the PI, the core group and volunteers would lead the development, implementation, and evaluation of all intervention events. Both peer leaders and the primary investigator will collaborate to develop specific events ("M-Groups"), guided by the findings in both the quantitative and qualitative studies. M-Groups will be held once every month. Events will be 2 hour activities focused on the aforementioned goals.
  Arms: MPowerment PrEP Promotion Intervention

SUMMARY:
The goal of the proposed research is to design a peer-based community intervention focused on addressing HIV stigma, and peer support to increase PrEP initiation in Prince George's County, MD. Participants will attend intervention events focused on stigma reduction and building community. Researchers will compare intervention and control group participants to see if there in a difference in PrEP initiation and adherence.

DETAILED DESCRIPTION:
Black gay, bisexual, and other Black sexual minority men (BSMM) are a priority population and experience the highest rate of new HIV infections in the United States. Maryland (MD) is an HIV epicenter and ranks 4th in AIDS cases nationally; the state has several hotspots of HIV and AIDS cases in geographically distinct areas, including urban, suburban, and rural settings. Prince George's (PG) County is a majority Black suburban county (63% Black) bordering Washington, DC, with the highest per capita income for Black people in the nation, yet the second highest incidence and prevalence of HIV in the DC greater metropolitan area. It is an understudied region in the "Ending the Epidemic" initiative to end HIV in the United States. Despite the availability of PrEP for prevention and overall economic resources in this area, uptake among BSMM remains low. Greater understanding of factors impacting PrEP utilization among BSMM in this population and region of the U.S. are necessary for successful HIV prevention for BSMM. Additionally, extant literature specific to PrEP use in PG county is extremely limited.

Internalized stigma is an important and understudied factor that can deter PrEP use among BSMM, similar to the well documented associations between internalized stigma and several HIV risk behaviors among SMM. Research has consistently shown the impact of stigma on several HIV-related outcomes among SMM, including HIV stigma that deters uptake of HIV prevention. In contrast, social support can facilitate HIV prevention behaviors. Internalized stigma and peer social support are potentially modifiable factors that may directly impact PrEP acceptability and PrEP stigma; the associations between internalized stigma and PrEP use are still notably understudied. Despite this, interventions promoting PrEP use have largely not addressed internalized stigma as a potential barrier to uptake.

The goal of the proposed research is to design a peer-based community intervention focused on addressing HIV stigma, HIV knowledge, and peer BSMM support to increase PrEP initiation in Prince George's County, MD. The investigators will adapt the MPowerment peer-based model: This is a CDC-developed evidence-based intervention originally designed to reduce sexual risk and improve peer support through the use of peer-led activities and discussions, often in a drop-in center. There have been several successful adaptations of the MPowerment model in different settings. The investigators are adapting the model to focus on improving PrEP initiation through focusing on peer support, and reducing internalized stigma, including HIV stigma, through peer-led events and activities. The following are our aims:

Aim 1. Using ethnographic methods (participant and direct observation), study peer-peer interactions/exchanges and HIV prevention communications in two ongoing MPowerment programs, one in Falls Church, VA (suburban) and the other in Washington, DC (urban).

Aim 2. Conduct 32 in depth interviews to inform adapting an MPowerment intervention to reduce internalized stigma and increase PrEP uptake among BSMM in PG County. This would inform intervention site selection, promotion materials, and design of events and activities.

Aim 3. Pilot test a community-based pretest-posttest intervention (n=130) to increase PrEP uptake in PG County, based on the MPowerment model, with a focus on reducing internalized HIV stigma and increasing social support and resilience.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Black
* HIV-negative
* 18 years of age or older
* Either residing in Prince George's County Maryland, or having a sexual partner in Prince George's County Maryland within the past year.

Exclusion Criteria

* HIV Positive
* Refusal of HIV testing

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a PreP prescription within one month of intervention completion. | Within 1 month of intervention completion.
  This is the number of participants who receive an initial prescription for Pre-exposure prophylaxis. Investigators will refer individuals participating in the intervention for PrEP use. Those who provide either a PrEP prescription, or a PrEP bottle with their prescription information, will be considered as initiating PrEP use.
Number of participants with a positive blood spot test for PrEP 6 months following the intervention. | 6 months post-intervention.
  6 months following the intervention completion, investigators will mail a blood spot collection kit to participants, with return postage. When mailed back, investigators will test the dried blood spots for the presence of PrEP using a chemistry analyzer. Those who test positive will be considered as "PrEP adherent".

CONTACTS AND LOCATIONS:
Overall Officials: Rodman Turpin, PhD, Principal Investigator — George Mason University
Locations (1):
- George Mason University, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
The investigators are still working on developing a plan for data dissemination.

REFERENCES:
- [Background] Sullivan PS, Mena L, Elopre L, Siegler AJ. Implementation Strategies to Increase PrEP Uptake in the South. Curr HIV/AIDS Rep. 2019 Aug;16(4):259-269. doi: 10.1007/s11904-019-00447-4. PMID 31177363
- [Background] Sun Z, Gu Q, Dai Y, Zou H, Agins B, Chen Q, Li P, Shen J, Yang Y, Jiang H. Increasing awareness of HIV pre-exposure prophylaxis (PrEP) and willingness to use HIV PrEP among men who have sex with men: a systematic review and meta-analysis of global data. J Int AIDS Soc. 2022 Mar;25(3):e25883. doi: 10.1002/jia2.25883. PMID 35255193
- [Background] Hillis A, Germain J, Hope V, McVeigh J, Van Hout MC. Pre-exposure Prophylaxis (PrEP) for HIV Prevention Among Men Who Have Sex with Men (MSM): A Scoping Review on PrEP Service Delivery and Programming. AIDS Behav. 2020 Nov;24(11):3056-3070. doi: 10.1007/s10461-020-02855-9. PMID 32274670
- [Background] Golub SA. PrEP Stigma: Implicit and Explicit Drivers of Disparity. Curr HIV/AIDS Rep. 2018 Apr;15(2):190-197. doi: 10.1007/s11904-018-0385-0. PMID 29460223
- [Background] Calabrese SK. Understanding, Contextualizing, and Addressing PrEP Stigma to Enhance PrEP Implementation. Curr HIV/AIDS Rep. 2020 Dec;17(6):579-588. doi: 10.1007/s11904-020-00533-y. Epub 2020 Sep 23. PMID 32965576
- [Background] Johnson J, Radix A, Copeland R, Chacon G. Building Racial and Gender Equity into a National PrEP Access Program. J Law Med Ethics. 2022;50(S1):55-59. doi: 10.1017/jme.2022.37. PMID 35902091
- [Background] Touger R, Wood BR. A Review of Telehealth Innovations for HIV Pre-Exposure Prophylaxis (PrEP). Curr HIV/AIDS Rep. 2019 Feb;16(1):113-119. doi: 10.1007/s11904-019-00430-z. PMID 30701404
- [Background] Dangerfield DT 2nd, Lipson A, Anderson JN. HIV PrEP Clinician Communication Preferences Among Black Sexual Minority Men. AIDS Educ Prev. 2022 Apr;34(2):168-181. doi: 10.1521/aeap.2022.34.2.168. PMID 35438541
- [Background] Bavinton BR, Grulich AE. HIV pre-exposure prophylaxis: scaling up for impact now and in the future. Lancet Public Health. 2021 Jul;6(7):e528-e533. doi: 10.1016/S2468-2667(21)00112-2. Epub 2021 Jun 2. PMID 34087117
- [Background] Sullivan PS, Siegler AJ. Getting pre-exposure prophylaxis (PrEP) to the people: opportunities, challenges and emerging models of PrEP implementation. Sex Health. 2018 Nov;15(6):522-527. doi: 10.1071/SH18103. PMID 30476461

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-14): https://cdn.clinicaltrials.gov/large-docs/08/NCT06141408/Prot_SAP_000.pdf